CLINICAL TRIAL: NCT07037615
Title: The Impact of Different Sedation Regimens on Hemodynamics in Patients Undergoing Mechanical Ventilation With Shock
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Li Shu, associate professor, Peking University People's Hospital
Other Study IDs: 2025-Z-44
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Mechanically Ventilated Patients With Shock
Keywords: Mechanically ventilated patients with shock; Sedation; Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cumulative vasoactive support duration <1 hour/24h: On day 28 after ICU admission, patients were assessed for vasoactive drug independence, defined as vasoactive drug infusion not exceeding 60 minutes within any continuous 24-hour window.
- Cumulative vasoactive support duration >1 hour/24h: On day 28 of ICU admission or thereafter, the patient underwent a vasoactive drug dependence assessment, defined as vasoactive drug infusion time exceeding 60 minutes within any continuous 24-hour window.

SUMMARY:
Mechanical ventilation is a common therapeutic intervention in the intensive care unit (ICU). However, patients undergoing mechanical ventilation often experience agitation, unplanned extubation, patient-ventilator asynchrony, and even neuroendocrine-immune dysregulation, sympathetic overexcitation, and organ dysfunction due to discomfort and pain. Sedation therapy mitigates patient stress, enhances comfort, and ensures the smooth implementation of mechanical ventilation, making it an essential component of treatment for ventilated patients. Nevertheless, sedation may impact peripheral vascular tone, leading to hemodynamic instability and exacerbating inadequate peripheral perfusion.

The precise implementation of sedation therapy to minimize adverse effects remains unclear. This prospective observational study will enroll critically ill patients with shock requiring mechanical ventilation. We will examine the effects of different sedation strategies-including sedation assessment protocols, sedative types, sedation duration, and daily awakening trials-on hemodynamics in this population. The study aims to explore optimized sedation regimens and provide evidence-based guidance for precision sedation therapy in clinical practice.

DETAILED DESCRIPTION:
Critically ill patients requiring mechanical ventilation in the ICU frequently present with concurrent shock. The hemodynamic effects of sedative agents may further exacerbate circulatory instability. Studies indicate that 34% of ICU patients require simultaneous mechanical ventilation and vasoactive agent support. Among ARDS patients, over 60% develop shock, with approximately 65% necessitating vasopressor administration.

Common sedatives like propofol and dexmedetomidine, despite being first-line choices, exhibit significant hemodynamic side effects:

* **Propofol** induces hypotension (incidence: 20%) through vasodilation, sympathetic suppression, and bradycardia.
* **Dexmedetomidine** causes hypotension and bradycardia at low doses, while triggering vasoconstriction via peripheral α-2 receptor activation at high doses-both scenarios reduce cardiac output.

Additional factors affecting hemodynamic stability include sedation depth, duration, and daily awakening protocols. Deep sedation may mask dynamic assessment of fluid responsiveness, delaying shock resuscitation. Conversely, daily awakening-though reducing ventilation duration-may increase circulatory fluctuations through stress responses. These complex interactions necessitate balancing sedation efficacy and circulatory stability in shock patients, yet standardized protocols for this population remain lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Receiving invasive mechanical ventilation, with endotracheal intubation -performed <12 hours before enrollment;
* Patient requiring sedative and analgesic medications;
* Hemodynamic instability: Hypotension (systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg) occurring within 6 hours before intubation to 6 hours after intubation, requiring continuous vasoactive medication therapy for >1 hour.

Exclusion Criteria:

* Pregnant or breastfeeding patients;
* Patients with confirmed or suspected acute primary brain pathology (e.g., traumatic brain injury, intracranial hemorrhage, stroke, hypoxic brain injury);
* Patients with confirmed or suspected spinal cord injury or other pathologies likely to cause permanent or prolonged weakness;
* Patients with known allergy to the analgesic, sedative, or vasoactive medications used in the study protocol;
* Patients receiving palliative care or with an expected survival of ≤48 hours; Patients previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
28-day vasoactive drug-free duration | The observation period commenced upon enrollment and continued for 7 days or until ICU discharge, whichever occurred first.

SECONDARY OUTCOMES:
Cumulative vasoactive drug dose during the first 7 days post-enrollment | The observation period commenced upon enrollment and continued for 7 days or until ICU discharge, whichever occurred first.
Incidence of new-onset organ failure (respiratory/circulatory/renal) within 7 days | The observation period commenced upon enrollment and continued for 7 days or until ICU discharge, whichever occurred first.
7-day sedation goal attainment rate | 7-day sedation goal attainment rate
28-day all-cause mortality | 28-day all-cause mortality
ICU-free days within 28 days | ICU-free days are calculated as 28 days minus the total number of days (or partial days) spent in the ICU. All patients who die before day 28 or prior to ICU discharge are assigned 0 ICU-free days.
Delirium duration within 28 days，Incidence of delirium | Delirium duration is defined as the number of days the patient was alive and had documented delirium. For patients discharged from the ICU before day 28, no further delirium assessments were conducted outside the ICU.
Ventilator-free days within 28 days | Ventilator-free days (VFDs) within 28 days are defined as the number of days the patient was alive and free from invasive mechanical ventilation for at least 48 consecutive hours (successful extubation).

CONTACTS AND LOCATIONS:
Overall Officials: Shu Li, doctor, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD，all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 1 years after publication
Access Criteria: The date used and/or analyzed during the current study are available from the investigator on reasonable request